CLINICAL TRIAL: NCT00014638
Title: Open Label, Multicenter Trial Of Femera (Letrozole) 2.5 mg As First-line Therapy In Postmenopausal Women With Metastatic Breast Cancer Relapsing Following Adjuvant Tamoxifen Therapy
Brief Title: Letrozole in Treating Postmenopausal Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000068583; NOVARTIS-CFEM345A-US10
Record Dates: First submitted 2001-04-10; First posted 2003-11-13 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

INTERVENTIONS:
Drug: letrozole

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of cancer cells. Letrozole may fight breast cancer by reducing the production of estrogen.

PURPOSE: Phase IV trial to study the effectiveness of letrozole in treating postmenopausal women who have metastatic breast cancer that has been previously treated with tamoxifen.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the time to progression of postmenopausal women with metastatic breast cancer treated with letrozole (Femara) as first-line therapy. II. Determine the objective response rate, time to treatment failure, survival rate, and changes in symptom distress in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified according to time to diagnosis of metastatic disease. Patients receive oral letrozole (Femara) daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 590 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of metastatic breast cancer Measurable or evaluable disease Postmenopausal No spontaneous menses for at least 5 years (including chemotherapy-induced amenorrhea) Spontaneous menses within the past 5 years allowed if amenorrheic for at least 12 months and LH and FSH in postmenopausal normal range (including chemotherapy-induced amenorrhea) Bilateral oophorectomy Radiotherapy castration and amenorrheic for at least 3 months Hormone receptor status: Estrogen-receptor (ER) and/or progesterone-receptor (PR) positive No ER and PR negative or unknown tumors

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: See Disease Characteristics Performance status: Karnofsky 50-100% WHO 0-2 Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Corrected serum calcium less than 11.6 mg/dL Other: No known hypersensitivity to any of the constituents of the study drug No history of noncompliance to medical regimens No unreliability Not pregnant or nursing Fertile patients must use effective contraception HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent anticancer immunotherapy or biological response modifiers Chemotherapy: See Disease Characteristics Prior adjuvant or neoadjuvant chemotherapy with adjuvant tamoxifen allowed No concurrent anticancer chemotherapy Endocrine therapy: See Chemotherapy No other concurrent anticancer endocrine therapy (including steroids) Radiotherapy: See Disease Characteristics No concurrent radiotherapy to sole site of disease Concurrent radiotherapy to a limited area (e.g., for painful disease) allowed Surgery: See Disease Characteristics No prior adrenalectomy or hypophysectomy Other: At least 30 days since prior systemic investigational drugs At least 7 days since prior topical investigational drugs No other concurrent investigational drugs Concurrent bisphosphonates (e.g., zoledronic acid) for bone metastasis allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-01; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Petrone, SCRS, Study Chair — Novartis Pharmaceuticals
Locations (20):
- United States (20):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Long Beach Memorial Breast Center, Long Beach, California
  - Cancer Research Network, Inc., Hollywood, Florida
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Pharm Research, Pinecrest, Florida
  - Cancer Research Network Inc., Plantation, Florida
  - Good Samaritan Medical Center, West Palm Beach, Florida
  - Illinois Oncology, Ltd., Belleville, Illinois
  - Joliet Oncology/Hematology Associates, Ltd., Joliet, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Southwest Oncology Association, Lafayette, Louisiana
  - New Mexico Oncology-Hematology, Albuquerque, New Mexico
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - Oncology Partnership Network, Cincinnati, Ohio
  - Memphis Cancer Center, Memphis, Tennessee
  - Dial Research Associates, Inc., Nashville, Tennessee
  - Center for Oncology Research and Treatment, Medical City Hospital, Dallas, Texas
  - Intermountain Hematology/Oncology Associates, Inc., Salt Lake City, Utah
  - Cascade Cancer Center, Kirkland, Washington